CLINICAL TRIAL: NCT06447987
Title: Phase Ib Study to Evaluate Humanized CD19-Specific CAR T Cells Following Lymphodepleting Chemotherapy in Adult Patients With Relapsed/Refractory CD19+ B-Cell Acute Lymphoblastic Leukemia
Brief Title: Humanized CD19-Specific CAR T Cells for the Treatment of Patients With Positive Relapsed or Refractory CD19 Positive B-Cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23328; NCI-2024-03338 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23328 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-05-09; First posted 2024-06-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Cetuximab; Cyclophosphamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (huCD19-CAR T) (Experimental): Patients undergo leukapheresis then receive lymphodepletion chemotherapy with fludarabine IV and cyclophosphamide IV on days -5, -4 and -3 and huCD19-CAR T IV cells over 10-15 minutes on day 0. Patients may optionally receive cetuximab IV over 60-120 minutes at least 28 days post T cell infusion and undergo alloHCT. Additionally, patients undergo ECHO or MUGA, CT or PET/CT and optional MRI on study and bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Biological: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes; Biological: Cetuximab; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo alloHCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Biological: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes — Given IV
  Other Names: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T Cells; CD19R(EQ)28zeta/EGFRt+ Naive and Memory T Cells; CD19R(EQ)28zetaEGFRt+ Tn/mem Cells
Biological: Cetuximab — Given IV
  Other Names: C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Procedure: Computed Tomography — Undergo CT and PET
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase Ib trial tests the safety, side effects, and effectiveness of humanized (hu)CD19-chimeric antigen receptor (CAR) T cell therapy in treating patients with CD19 positive B-cell acute lymphoblastic leukemia (ALL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). CAR T-cell therapy is a treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein, such as CD19, on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the huCD19 positive CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Chemotherapy drugs, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. huCD19-CAR T cell therapy may be safe, tolerable and effective in treating patients with relapsed or refractory CD19 positive ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of Tn/mem-enriched huCD19(VH4VK1)(dCH2)BBzeta/EGFRt+ T cells (huCD19 CAR T) as single-dose monotherapy by evaluation of toxicities including type, frequency, severity, attribution, time course and duration.

II. Determine the maximum feasible dose (MFD)/recommended phase 2 dose(s) schedule (RP2D) of huCD19 CAR T as single-dose monotherapy on relapsed/refractory (r/r) ALL patients.

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates of complete remission (complete remission [CR] /complete response with incomplete bone marrow recovery [CRi]) rate(s).

II. Overall response rate (CR, CRi): best response. III. Duration of response (CR, CRi). IV. Minimal residual disease (MRD)- negative CR/CRi. V. The number and rate of bridging to transplant. VI. Estimate the progression free survival (PFS) and overall survival (OS) rate, at 6-months and 1-year post (first) huCD19 CAR T cell infusion.

EXPLORATORY OBJECTIVES:

I. Access the expansion and persistence of T cell via flow cytometry in blood, bone marrow (BM) and cerebrospinal fluid (CSF).

II. Assess the phenotype and activation status of CAR T via flow cytometry, polymerase chain reaction (PCR), and cytokine analysis.

III. Assess CAR T cell clonal expansion and repertoires of endogenous T cells. IV. Assess immunophenotyping and functional analyses of CAR T cell products. V. Determine the role of the immunologic milieu. VI. Evaluation of B cell aplasia. VII. Serum cytokine measurement. VIII. Tumor antigen analysis. XIV. Evaluation of Immunogenicity by enzyme-linked immunosorbent assay (ELISA). X. For subjects who receive cetuximab for CAR T cell ablation, assess the activity of infusional cetuximab to eliminate transferred huCD19-CAR T cells.

OUTLINE: This is a dose-escalation study of huCD19-CAR T, followed by a dose-expansion study.

Patients undergo leukapheresis then receive lymphodepletion chemotherapy with fludarabine ntravenously (IV) and cyclophosphamide IV on days -5, -4 and -3 and huCD19-CAR T IV cells over 10-15 minutes on day 0. Patients may optionally receive cetuximab IV over 60-120 minutes at least 28 days post T cell infusion and undergo allogeneic hematopoietic cell transplantation (alloHCT). Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan ((MUGA), computed tomography (CT) or positron emission tomography (PET)/CT and optional magnetic resonance imaging (MRI) on study and bone marrow biopsy and aspiration and blood sample collection throughout the study.

After completion of study treatment, patients are followed up monthly for 1 year then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
  * Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed. However, the research participant is allowed to proceed with lymphodepletion and T cell infusion only after the translated full consent form is signed
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) 0-2 / Karnofsky performance status (KPS) ≥ 70
* Histologically confirmed CD19+ relapsed/refractory ALL with at least 2 prior lines of therapy

  * Prior alloHCT > 100 days prior to enrollment may be considered a prior line of therapy
* Research participants with confirmed 1st or higher relapse of disease by morphology, cytogenetics or molecular, or research participants with refractory or residual disease

  * Participants with central nervous system (CNS) involvement by leukemia (CNS2 and CNS3) may be considered eligible after discussions with the study team
  * Patients with only MRD+ disease may be eligible
  * Patients with isolated extramedullary disease may also be eligible
* Total bilirubin ≤ 2.0 X upper limit of normal (ULN) (unless has Gilbert's disease or related to leukemia involving the liver)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN (unless related to leukemia involving the liver)
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN (unless related to leukemia involving the liver)
* Creatinine clearance of ≥ 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula
* Left ventricular ejection fraction (LVEF) ≥ 45%

  * Note: To be performed within 28 days prior to start of protocol therapy
* Cardiac function (12 lead-electrocardiogram [ECG]): Corrected QT interval (QTc) must be ≤ 480 msec
* Oxygen (O2) saturation > 92% on room air

  * Note To be performed within 28 days prior to start of protocol therapy
* Seronegative for HIV quantitative polymerase chain reaction (qPCR), hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed. OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. The viral load must be undetectable
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to start of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* ELIGIBILITY TO PROCEED WITH PERIPHERAL BLOOD MONONUCLEAR CELLS (PBMC) COLLECTION FOR CAR T CELL MANUFACTURING
* Research participant has signed the 'screening and leukapheresis' informed consent
* Research participant must have appropriate venous access, have a central line or be willing to undergo central or temporary line placement
* The last dose of systemic chemotherapy must be at least 2 weeks before the leukapheresis procedure with the following exceptions:

  * Steroids and vincristine are allowed up to 7 days prior to leukapheresis.
  * Intrathecal chemotherapy is allowed up to 3 days prior to leukapheresis.
  * Tyrosine kinase inhibitors are allowed up to 48 hours prior to leukapheresis.
  * Hydrea is allowed up to 48 hours prior to leukapheresis.
  * The research participant cannot be on ≥ 7.5 mg prednisone or equivalent doses of other corticosteroids at the time of leukapheresis. Note: Topical and inhaled corticosteroids in standard doses and physiologic replacement for subjects with adrenal insufficiency are allowed
* The last dose of prior targeted agents, immunotherapy or radiation must be at least 2 weeks before the leukapheresis procedure
* If the research participant has undergone prior alloHCT, 100 days must have elapsed since allogeneic stem cell transplant to undergo PBMC collection for CAR T cell manufacturing
* ELIGIBILITY TO UNDERGO LYMPHODEPLETION
* Research participant's absolute leukemic blast count does not exceed 10,000 cells/uL
* The last dose of chemotherapy, maintenance therapy, radiation therapy, biological therapy, and/or immunotherapy must have been 7 days prior to start of lymphodepletion
* The following washout periods must be met:

  * Corticosteroids 3 days
  * Biologic agents 3 half lives
  * Oral chemotherapeutic agents 3 half lives
  * Intrathecal chemotherapy 3 days
  * Chemo and/or immunotherapy 2 weeks
  * Local radiation to sites 7 days
  * Non myeloablative agents 7 days
  * Investigational agents 2 weeks, or at least 3 half lives
  * Hydroxyurea no washout period
* Research participant has a released cryopreserved CAR T cell product for CAR T cell infusion on approximately day 0 (performed no more than 7 days prior to start of lymphodepletion)
* ECOG < 2 / KPS ≥ 70 (performed no more than 7 days prior to start of lymphodepletion)
* No ongoing post treatment ≥ grade 3 non-heme toxicities (with exception of grade 3 glucose intolerance, cholesterol, triglyceride, peripheral neuropathy, and hyperglycemia) (performed no more than 7 days prior to start of lymphodepletion)
* Research participant does not require supplemental oxygen to keep saturation greater than or equal to 92% and/or does not have any radiographic abnormalities on chest x-ray that are progressive (performed no more than 7 days prior to start of lymphodepletion)
* Research participant does not require pressor support and/or does not have symptomatic cardiac arrhythmias (performed no more than 7 days prior to start of lymphodepletion)
* Research participant does not have a fever exceeding 38.5 degree Celsius (C); there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to lymphodepletion and/or there aren't any indications of meningitis (performed no more than 7 days prior to start of lymphodepletion)
* Research participant serum total bilirubin does not exceed 2.5X normal limit or transaminases do not exceed 3X normal limit unless related to underlying leukemia (to be discussed at the discretion of the PI/study team) (performed no more than 7 days prior to start of lymphodepletion)

  * Note: in the event a participant has elevated levels of liver enzymes possibly related to underlying disease/disease progression, the participant will still be considered eligible
* Research participant serum creatinine ≤ 2 mg/dL (performed no more than 7 days prior to start of lymphodepletion)
* Research participant does not have uncontrolled seizure activity (performed no more than 7 days prior to start of lymphodepletion)
* ELIGIBILITY TO PROCEED WITH CAR T CELL INFUSION
* No ongoing post treatment ≥ grade 3 non-heme toxicities (with exception of grade 3 glucose intolerance, cholesterol, triglyceride, peripheral neuropathy, and hyperglycemia)
* Prednisone (or prednisone equivalent) dose of ≤ 7.5 mg/kg/day is allowed
* Prohibited medications have not been administered
* KPS ≥ 70
* No untreated or active systemic infection
* No Class III/IV cardiovascular disability according to the NYHA Classification
* Research participant does not require supplemental oxygen to keep saturation greater than or equal to 92% and/or does not have any radiographic abnormalities on chest x-ray that are progressive
* Research participant does not require pressor support and/or does not have symptomatic cardiac arrhythmias
* Research participant does not have a fever exceeding 38.5 degree C; there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to T cell infusion and/or there aren't any indications of meningitis
* Research participant serum total bilirubin does not exceed 2.5X normal limit or transaminases do not exceed 3X normal limit unless related to underlying leukemia (to be discussed at the discretion of the PI/study team)
* Research participant serum creatinine ≤ 2 mg/dL
* Research participant does not have uncontrolled seizure activity
* ELIGIBILITY TO PROCEED WITH OPTIONAL CAR T CELL ABLATION
* Research participant has > 1% CAR T cells in the peripheral blood
* No known hypersensitivity to cetuximab
* Not requiring supplemental oxygen or mechanical ventilation, oxygen saturation 92% or higher on room air
* Not requiring pressor support, no symptomatic cardiac arrhythmias, no acute coronary syndrome, or uncontrolled hypertension
* Serum creatinine did NOT increase by more than 2.5 fold from base line (at time of screening )
* Adequate liver function defined as total bilirubin < 3.0 mg/dl, AST < 5 x ULN; ALT < 5 x ULN
* Research participant without clinically significant encephalopathy/new focal deficits
* No clinical evidence of uncontrolled active infectious process

Exclusion Criteria:

* Allogeneic stem cell transplant within 100 days at the time of enrollment
* Received prior CAR T therapy within 90 days of enrollment

  * EXCEPTION: Participants who have previously received B-cell-activating factor receptor (BAFFR)-CAR T cells will be excluded from this study
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent(s)
* History or presence of clinically relevant CNS pathology such as uncontrolled seizure disorder, recent stroke, severe brain injuries, dementia, cerebellar disease or psychosis
* Autoimmune disease or active graft versus host disease (GVHD) requiring systemic immunosuppressant therapy
* Class III/IV cardiovascular disability according to the New York Heart Association (NYHA) Classification
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for ≥ 2 years
* Clinically significant uncontrolled illness
* Active systemic uncontrolled infection requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection

  * Subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded

    * Subjects who are hepatitis B core antibody positive (or have a known history of HBV infection) should be monitored quarterly with a quantitative PCR test for HBV deoxyribonucleic acid (DNA). HBV monitoring should last until 12 months after the last dose of study drug. Any subject with a rising viral load (above lower limit of detection) should discontinue study drug and have antiviral therapy instituted and a consultation with a physician with expertise in managing hepatitis B. Subjects who are core antibody (Ab) positive at study enrollment are strongly recommended to start Entecavir before start and until completion of study treatment
    * Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded
* Females only: Pregnant or breastfeeding
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of topical or inhaled steroids is not exclusionary. Physiologic replacement of steroids (prednisone ≤ 7.5 mg /day or equivalent) is allowed
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 28 days after T cell infusion
  Toxicity/ adverse events will be graded using Common Terminology Criteria for Adverse Events version 5.0. Cytokine release syndrome and neurotoxicity will be graded using American Society for Transplantation and Cellular Therapy Consensus Criteria. Toxicity will be summarized and tabulated by count and percentage of subjects stratified by severity (grade), relatedness, terms or organ level.

SECONDARY OUTCOMES:
Percentage of patients undergoing leukapheresis who get sufficient T cells manufactured and infused at assigned dose level | At time of infusion
Overall response rate (ORR) | Up to 28 days post infusion
  ORR will be defined as the percentage of subjects who experience a best response of either complete response (CR) or complete response with incomplete bone marrow recovery (CRi). Exact 95% confidence intervals will be calculated.
Progression-free survival (PFS) | From the start of CD-19 CAR T cell infusion to the date of death or disease progression/relapse, whichever occurring first, assessed up to 15 years
  PFS over time will be assessed by Kaplan-Meier method.
Duration of response (DOR) | From the start of CD19-CAR T cell infusion to the date of death or disease progression/relapse, whichever occurring first, assessed up to 15 years
  DOR will be defined as the time from the first achievement of CR or CRi after infusion through disease relapse or progression or death.
Overall survival (OS) | From start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 15 years
  OS over time will be assessed by Kaplan-Meier method.
Minimal residual disease (MRD) | Up to 2 years post infusion
  MRD relapse will be defied as detectable of leukemic cells at > 0.01% in morphological remission bone marrow.
Extramedullary relapse | Up to 2 years post infusion
  Extramedullary relapse will be defined as documented relapse outside the bone marrow.
Transplant OS | At days 30 and 100, 6 months, and years 1 and 2 post alloHCT
  Transplant OS will be defined as the duration of time from start of allogeneic hematopoietic cell transplant (alloHCT) to time of death (due to any cause). OS over time will be assessed by Kaplan-Meier method.
Transplant PFS | At days 30 and 100, 6 months, and years 1 and 2 post alloHCT
  Transplant PFS will be defined as the duration of time from start of alloHCT treatment to time of progression or death, whichever comes first. PFS over time will be assessed by Kaplan-Meier method.
Transplant relapse/progression | At days 30 and 100, 6 months, and years 1 and 2 post alloHCT
Non-relapse mortality (NRM) | At days 30 and 100, 6 months, and years 1 and 2 post alloHCT
  NRM will be defined as death occurring in a patient from causes other than relapse or progression. NRM will be measured from start of treatment until non-disease related death or last follow up, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Aldoss, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States